CLINICAL TRIAL: NCT05035472
Title: Comparison of the Potency of Prophylactic Norepinephrine and Phenylephrine Boluses for Postspinal Anesthesia Hypotension in Patients With Severe Preeclampsia During Caesarean Section
Brief Title: The Potency of Prophylactic Norepinephrine and Phenylephrine Boluses for Postspinal Anesthesia Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2021-3
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Adverse Effect
Keywords: Norepinephrine; Phenylephrine; Postspinal anesthesia hypotension; Preeclampsia; Cesarean section
MeSH Terms: conditions — Pre-Eclampsia | interventions — Phenylephrine; Vasoconstrictor Agents; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylephrine group (Active Comparator): Prophylactic phenylephrine bolus simultaneous with spinal anesthesia
  Interventions: Drug: Phenylephrine
- Norepinephrine group (Experimental): Prophylactic norepinephrine bolus simultaneous with spinal anesthesia
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — An initial prophylactic bolus dose of phenylephrine (37.5μg) simultaneous with spinal anesthesia. If the patient did not respond adequately to the current dose (SBP decreased to < 80% of baseline), the dose was considered to have failed and the subsequent dose for the following patient was increased to the next higher dose level. The dose administered to subsequent patients varied by increments or decrements of 12.5 μg according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Vasopressors
  Arms: Phenylephrine group
Drug: Norepinephrine — An initial prophylactic bolus dose of norepinephrine (3μg) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 1 μg according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Vasopressors
  Arms: Norepinephrine group

SUMMARY:
The purpose of this study is to investigate the potency between prophylactic norepinephrine and phenylephrine boluses for postspinal anesthesia hypotension in patients with severe preeclampsia during caesarean section.

DETAILED DESCRIPTION:
Preeclampsia, which affects 5% to 7% of patients, is a significant cause of maternal and neonatal morbidity and mortality. Because of constricted myometrial spiral arteries with exaggerated vasomotor responsiveness, though blood pressure in patients with preeclampsia are apparently higher than healthy patients, placental hypoperfusion is more common. Spinal anesthesia is still the preferred mode of anesthesia in patients with preeclampsia for cesarean section. In preeclampsia patients, spinal anesthesia improve intervillous blood flow (provided that hypotension is avoided) which contribute to increase placental perfusion. Even so, 17-26% patients with preeclampsia experienced postspinal anesthesia hypotension due to the extensive sympathetic block that occurred with spinal anesthesia. As a potential substitute drug for phenylephrine and ephedrine, norepinephrine has gained traction for use in patients undergoing cesarean section. However, the ED50 (prevent postspinal hypotension in 50% of patients) and ED90 of prophylactic norepinephrine bolus is still unknown. The purpose of this study is to investigate the potency between prophylactic norepinephrine and phenylephrine boluses for postspinal anesthesia hypotension in patients with severe preeclampsia during caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥32 weeks
* American Society of Anesthesiologists physical status classification II to III
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Baseline blood pressure ≥180 mmHg
* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The dose that would be effective in preventing postspinal anesthesia hypotension in 50% (effective dose, ED 50) and 90% (ED90) of patients | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, Dr., Study Chair — General Hospital of Ningxia Medical University